CLINICAL TRIAL: NCT00326326
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study To Evaluate The Effect Of CP-778,875 On HDL-Cholesterol In Adult Subjects With Dyslipidemia And Type 2 Diabetes Mellitus
Brief Title: Effect of CP-778,875 on HDL-C in Subjects With Abnormal Lipid Levels and Type 2 Diabetes.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5561005
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Last update posted 2009-05-07 (Estimated); Status verified 2009-05

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

INTERVENTIONS:
Drug: CP-778,875

SUMMARY:
To assess the effect of CP-778,875 on HDL-C cholesterol in adult subjects with dyslipidemia and type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* HDL-C < or = 45 mg/dL for men and < or = 55 mg/dL for women
* Triglycerides between 150-500 mg/dL
* Fasting Plasma Glucose 140-240 mg/dL

Exclusion Criteria:

* Known cardiovascular, carotid, or peripheral vascular disease

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84
Dates: Start 2006-07; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
HDL-C Safety and Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- United States (29):
  - Pfizer Investigational Site, Anniston, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Greenbrae, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, DeFuniak Springs, Florida
  - Pfizer Investigational Site, Destin, Florida
  - Pfizer Investigational Site, Jupiter, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Conyers, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Mount Vernon, New York
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Bryan, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Newport News, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Yakima, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5561005&StudyName=Effect%20of%20CP-778%2C875%20on%20HDL-C%20in%20subjects%20with%20abnormal%20lipid%20levels%20and%20type%202%20diabetes.